CLINICAL TRIAL: NCT02669212
Title: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Brief Title: Myalgic Encephalomyelitis Chronic Fatigue at the National Institutes of Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 160058; 16-N-0058
Record Dates: First submitted 2016-01-29; First posted 2016-02-01 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-06-10

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome; Lyme Disease; Healthy Volunteers; Movement Disorder
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Lyme Disease; Movement Disorders | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteer Participants (Other): Healthy volunteer participants
  Interventions: Behavioral: Cardiopulmonary Exercise Test (CPET)
- ME/CFS Participants (Other): Participants with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
  Interventions: Behavioral: Cardiopulmonary Exercise Test (CPET)

INTERVENTIONS:
Behavioral: Cardiopulmonary Exercise Test (CPET) — All participants will undergo an exercise stress test

SUMMARY:
Background:

Post-Infectious Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (PI-ME/CFS) refers to long-lasting and disabling fatigue or malaise, inability to recover after exercise, and physical and emotional discomfort that may occur after a person has an infection. Researchers want to learn more about its causes.

Objective:

To learn more about PI-ME/CFS.

Eligibility:

Adults ages 18-60 years who have finished at least 7th grade education and either:

have ME/CFS that started after an infection

OR had Lyme disease, were treated, and returned to normal health

OR are healthy volunteers

Design:

Participants will initially have a 2-5 day inpatient visit at the National Institutes of Health Clinical Center in Bethesda. During the visit, participants will have:

Medical history

Physical exam

Intravenous (IV) line. A thin plastic tube is inserted into a vein.

Blood and urine collected

Magnetic resonance imaging (MRI). Participants will lie in a machine that takes pictures of their brain. They may get a dye through their IV.

Grip strength tested

Saliva, cheek swab, and stool collected

Tilt table test with measures of body functions such as sweating and breathing, blood pressure, and heart rate and blood and urine sample collection

Collection of blood cells. Participants can choose to have the blood drawn through the IV or through a machine that filters blood cells and returns the liquid blood back into the participant s vein.

Lumbar puncture. Fluid will be removed by placement of a needle between the back bones.

Heart monitoring

Sleep study for participants with PI ME/CFS

Questions about the participant s life and how they are feeling

Questions from a neuropsychologist

Questions from an occupational therapist for participants with PI ME/CFS

Questinos from a nutritionist

After the initial visit participants will return home. Participants evaluated for PI-ME/CFS during the first visit will have their information reviewed by an adjudication panel of experts in the diagnosis and care of ME/CFS to determine if they are eligible to participate in the second study visit.

Eligible participants will be invited back for a second study visit. If a participant was taking certain medications during the first visit, they may be asked to taper off of them prior to the second visit and report any problems. They will also receive an activity monitor, fatigue diary, and nutrition log to use for at least one week prior to their second visit.

Participants who are eligible will return for a 5-10 day inpatient hospital visit at the National Institutes of Health Clinical Center. During the visit, participants will undergo measurements before and up to 96 hours after performing a stationary bike exercise test. The purpose of the exercise test is to provoke ME/CFS symptoms (post-exertional malaise). Tests will be performed before and after exercise testing. These include:

Sleeping in a room that measures how the body uses energy with EEG monitoring

Eating a controlled diet

Performing vigorous exercise for 10-15 minutes

Questions about how participants are feeling

Questions about what participants usually eat

Samples of saliva, blood, urine and stool

Wearing an activity monitor

Having an Xray that measures body composition

Thinking and memory tests

Heart monitoring

Transcranial magnetic stimulation. A brief electrical current to the scalp creates a magnetic pulse that affects brain activity.

Magnetic resonance imaging (MRI). Participants will lie in a machine that takes pictures of their brain. They will do thinking and exercise tasks during the MRI.

Lumbar puncture. Fluid will be removed by placement of a needle between the back bones.

DETAILED DESCRIPTION:
Objective:

The primary objective is to explore the clinical and biological phenotypes of post-infectious myalgic encephalomyelitis/chronic fatigue syndrome (PI-ME/CFS). The secondary objective is to explore the pathophysiology of fatigue and post-exertional malaise (PEM).

Study population:

Up to 206 persons will be enrolled as part of this protocol. Up to 150 persons aged 18-60 will be part of 3 study groups: 50 ME/CFS patients whose fatigue began after an infection, 50 non-fatigued participants with a documented history of a full recovery from COVID-19 infection, and 50 healthy volunteers. The study has a target of completing all study procedures on 20 enrolled participants in each group. Up to an additional 36 persons reporting a community diagnosis of ME/CFS will be enrolled into focus groups to discuss the experience of post-exertional malaise. Up to an additional 10 healthy volunteers and 10 ME/CFS patients may be enrolled to refine the protocol's electrophysiological and neuroimaging techniques.

Design:

This is a single-center, exploratory, cross-sectional study of PI-ME/CFS. Participants will have a phenotyping visit, which will encompass a 2-5 day long inpatient admission at the NIH Clinical Center. Case status for ME/CFS participants will be determined after the phenotyping visit by a case adjudication process utilizing an expert physician committee and published guidelines. Adjudicated participants meeting inclusion criteria will be invited back to participate in an exercise stress visit, which will encompass a 5-10 day long inpatient admission. Detailed subjective and objective measurements and biological specimens will be serially collected before and up to 96 hours after a peak exercise test capable of inducing post-exertional malaise during this visit. All procedures will be completed on all three study groups to allow for optimal inter-group comparisons.

Outcome measures:

The primary purpose of this protocol is to perform exploratory analysis of collected samples for the generation of new hypotheses regarding ME/CFS. The types of analyses to be performed will be wide ranging. Planned areas of focus include:

1. Characterization of the immune system and inflammation at baseline
2. Characterization of the pattern of microbiome in collected samples at baseline
3. Characterization of bioenergetics, autonomic, and metabolic function in collected samples at baseline
4. Characterization of neurocognition at baseline
5. Characterization of autonomic function at baseline

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusion criteria for all participants

  1. Adult participants aged 18-60 years at the time of enrollment.
  2. Self-reported completion of at least the 7th grade of school.
  3. Ability to speak, read, and understand English.
  4. Willing and able to complete all study procedures
  5. Participant has a primary care physician at the time of enrollment.
  6. Able to provide informed consent.
* Additional inclusion criteria for participants with PI-ME/CFS for the phenotyping visit:

  1. A self-reported illness narrative of the development of persistent fatigue and post-exertional malaise as the consequence of an acute infection. The persistent fatigue may have an acute onset or become progressively worse over 6 months.
  2. Licensed Independent Practitioner documentation of ME/CFS onset:

     * Medical documentation of absence of symptoms within one year of ME/CFS onset. This may include medical records, letters, or information gathered from telephone calls with study personnel.
     * Documentation of a medical evaluation for symptoms of an acute infection or documentation of a medical evaluation of persistent symptoms within 2 months following an assumed infection.
  3. Persistent fatigue and PEM onset less than 5 years prior to enrollment.
* Additional inclusion criteria for participants with PI-ME/CFS for the exercise stress visit:

  1. Be unanimously considered to be a case of PI-ME/CFS by the protocol s adjudication committee.
  2. Meet the 1994 Fukuda Criteria or the 2003 Canadian Consensus Criteria for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome or the Institute of Medicine Diagnostic Criteria..
  3. Have moderate to severe clinical symptom severity:

     * Severe fatigue as determined using the Multidimensional Fatigue Inventory (MFI): score of greater than or equal to 13 on the general fatigue subscale or greater than or equal to 10 on the reduced activity subscale.
     * Functional impairment as determined using the Short-Form 36 (SF-36): score of less than or equal to 70 physical function subscale, or less than or equal to 50 on role physical subscale, or less than or equal to 75 on social function subscale
* Additional inclusion criteria for healthy volunteer group:

None

* Additional inclusion criteria for COVID-19 Healthy Volunteers: documented prior COVID19 infection as evidenced by:

  1. A history of clinical manifestations compatible with COVID-19
  2. Laboratory evidence of Covid-19 infection:

     * Detectionof SARS-CoV-2RNA or antigen in nasopharyngeal swab, sputum, other sample source with Emergency Use Authorization/approval from the FDA; OR
     * A positive antibody test using an assay that has received Emergency Use Authorization/approval from the FDA
  3. Has been recovered from the COVID-19 infection for at least six months and no more than five years.

     EXCLUSION CRITERIA:
* Exclusion criteria for all participants:

  1. Current or past psychotic disorder including depression with psychosis, bipolar disorder, and schizophrenia
  2. Current DSM-5-defined major depression disorder, generalized anxiety disorder, post-traumatic stress disorder, panic disorder, or obsessive-compulsive disorder unless managed for more than six months with a stable treatment regimen
  3. Current or prior substance use disorder as diagnosed on the Structured Clinical Interview for DSM-5 (SCID-5).
  4. Current suicidal ideation
  5. History of head injury with loss of consciousness or amnesia lasting greater than a few seconds within lasta five years or lasting greater than 5 minutes at any point during their lifetime. Persons with medical record evidence of post-concussive symptoms lasting more than six months are also excluded.

     Persons with medical record evidence of post-concussive symptoms lasting more than six months are also excluded.
  6. Women who are pregnant, actively seeking to become pregnant, or have been pregnant in the year prior to study enrollment.
  7. Current or previous malignancy. Certain dermatologic malignancies (e.g. basal cell carcinoma) will be allowed. A history of malignancy that have fully resolved with surgical resection only (i.e. no chemotherapy, radiation therapy, or immunotherapy) will be allowed.
  8. Current systemic immunologic disorder (e.g. Type 1 diabetes, rheumatoid arthritis) will be excluded. Allergies requiring anti-histamines may not be an exclusion, but allergies requiring immunosuppressants may be an exclusion.
  9. Current or previous long term immune suppressive or immunomodulatory therapy. Systemic steroid use, even short-term, must not have been used within the month prior to enrollment
  10. Any medical condition (eg, congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, severe osteoarthritis, poorly controlled asthma) that would make the study procedures risky for the participant (e.g. exercise-induced angina and asthma) or that may confound the study results (e.g. untreated obstructive sleep apnea, severe osteoarthritis).
  11. Participation in a clinical protocol (e.g. anti-inflammatory drug intervention study) which includes an intervention that may affect the results of the current study.
  12. Inability to perform the bicycling exercise task.
  13. Clinically significant claustrophobia
  14. Not willing to allow for research samples to be shared with other researchers.
  15. Employees or staff at NIH that are directly supervised by the primary investigator or associate investigators.
* Additional exclusion criteria for participants with PI-ME/CFS for phenotyping visit:

  1. Significant neurological disorder (e.g. neurodegenerative disorder, stroke, epilepsy).
  2. PI-ME/CFS disease severity that makes it impossible for the volunteer to leave the home or requires inpatient treatment.
  3. Suspected, probable, or confirmed Lyme disease per 2011 CDC Lyme Disease National Surveillance Case Definitions.
  4. Underlying illness that may cause fatigue such as thyroid dysfunction, hepatitis, or other systemic diseases.
* Additional exclusion criteria for participants with PI-ME/CFS for exercise stress visit:

  1. Current (within 1 week) use of prescription or over-the-counter medications, herbal supplements, or nutraceuticals that may influence brain excitability that the potential participant is either unwilling or clinically unable to safely wean off for the duration of the period of the exercise stress visit. The possibility for a potential participant to be weaned off medication will be cooperatively determined by both the clinical investigative team and personal physicians. Examples of medications that influence brain excitability include tricyclic antidepressants, hypnotic, antiepileptic, antipsychotic medication, stimulants, antihistamines, muscle relaxants, dopaminergic medications, and sleep medications.
* Additional exclusion criteria for healthy volunteer group:

  1. Substantial daily fatigue as determined using PROMIS-SF Fatigue: score of > 17.
  2. Significant neurological disorder (e.g. neurodegenerative disorder, stroke, epilepsy).
  3. Current (within 1 week) use of prescription or over-the-counter medications, herbal supplements, or nutraceuticals that may influence brain excitability
* Additional exclusion criteria for COVID-19 healthy volunteer group:

  1. Substantial daily fatigue as determined using PROMIS-SF Fatigue: score of >17.
  2. Significant neurological disorder (e.g. neurodegenerative disorder, stroke, epilepsy).
  3. Current (within 1 week) use of prescription or over-the-counter medications, herbal supplements, or nutraceuticals that may influence brain excitability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-N-0058.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were either referred to study investigators by their primary care physician or were self-referred either through the Patient Recruitment and Public Liaison (PRPL) office or direct contact. Interested participants were contacted by telephone to evaluate eligibility. Eligible participants were subsequently seen at the NIH Clinical Center for study visits. Recruitment began February 2016 and ended February 2020.
Pre-assignment Details: Participants underwent telephone screening followed by a medical record review/discussion with the participant's physician to determine general eligibility. Participants were invited to campus to determine if they met inclusion/exclusion criteria for the phenotyping phase of the study. After the phenotyping visit, results were reviewed by a panel of expert adjudicators to determine case status and eligibility for the exercise phase of the protocol. No Lyme disease participants were recruited.
Groups:
- Healthy Volunteer Participants: Participants found to be healthy after a medical and psychiatric evaluation.
Period: Overall Study
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Started | 25 | 27
Completed | 21 | 17
Not Completed | 4 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Medical Condition | 3 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Excluded - determined NOT post-infectious | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.24 (13.46) | 37.82 (14.72) | 40.35 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 21 | 25 | 46
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cardiopulmonary Exercise Test (CPET) - ATVO2rel
Description: The Relative Volume of Oxygen at the Anaerobic Threshold (ATVO2rel) was determined during a cardiopulmonary exercise test (CPET). ATVO2rel represents the volume of oxygen being consumed when a participant reaches AT, adjusted for their weight during the CPET. Results compared Healthy Volunteer Participants to ME/CFS Participants.
Time Frame: At time of AT during CPET
Population: COVID-19 pandemic halted return visit for participation in Exercise Phase of trial.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Healthy Volunteers: Participants found to be healthy after a medical and psychiatric evaluation who completed the Cardiopulmonary Exercise Test (CPET).
- ME/CFS Participants: ME/CFS Participants who complete the Cardiopulmonary Exercise Test (CPET)
Arm/Group | Healthy Volunteers | ME/CFS Participants
Number analyzed (Participants) | 9 | 9
mL/kg/min | 16.0 (4.3) | 10.6 (3.8)

2. Primary Outcome: Cardiopulmonary Exercise Test (CPET) - RER
Description: The Respiratory Exchange Ratio (VCO2/VO2) was determined during a cardiopulmonary exercise test (CPET). VCO2/VO2 is calculated by measuring the volume of carbon dioxide and oxygen the participant breathes during CPET. When the volume of carbon dioxide exceeds that of oxygen, it reflects a change from aerobic metabolism to anaerobic metabolism. When a participant has a Respiratory Exchange Ratio (RER) during CPET that is equal or greater than 1.1 it is considered a sufficient exercise effort. Results compared Healthy Volunteer Participants to ME/CFS Participants.
Time Frame: At time of AT during CPET
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Healthy Volunteer Participants: Participants found to be healthy after a medical and psychiatric evaluation who completed the Cardiopulmonary Exercise Test (CPET).
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 9 | 9
Ratio | 1.3011 (0.0791) | 1.2415 (0.1156)

3. Other Pre Specified Outcome: Characterization of Total Body Energy Use (Bioenergetics/Metabolic)
Description: The total amount of energy expended per unit of time as measured by whole-room indirect calorimetry. This method measures the amount of oxygen consumed and carbon dioxide produced which can be used to calculate the amount of energy produced by biological oxidation and is measured by kilocalories per day. Measures were taken from Healthy and ME/CFS participants.
Time Frame: 12 hours
Population: Procedure added to Phenotyping Phase after enrollment started.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 11 | 16
kcal/day | 1858.9 (353.3) | 1862.1 (390.5)

4. Other Pre Specified Outcome: Characterization of the Immune System and Inflammation - WBC
Description: Blood and CSF were collected from healthy and ME/CFS participants at baseline. A comparison of the White Blood Cell (WBC) Count, i.e., a measurement of the number of white blood cells in the blood, in the two populations is reported. Low values can suggest immune deficiencies. High values can suggest infection or inflammation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: number of WBCs(K)/uL
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 21 | 17
number of WBCs(K)/uL | 5.907 (1.536) | 6.143 (1.243)

5. Other Pre Specified Outcome: Characterization of the Immune System and Inflammation - ESR
Description: Blood and CSF were collected from healthy and ME/CFS participants at baseline. A comparison of the results of the Erythrocyte Sedimentation Rate (ESR), i.e., a measure of how quickly red blood cells settle at the bottom of a test tube, in the two populations is reported. A faster than normal rate of settling suggests inflammation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 21 | 17
mm/hr | 7.43 (6.13) | 10.1 (11.9)

6. Other Pre Specified Outcome: Characterization of the Immune System and Inflammation - CRP
Description: Blood and CSF were collected from healthy and ME/CFS participants at baseline. A comparison of the results of C-Reactive Protein (CRP), i.e., a measurement of a protein that is made by the liver, in the two populations is reported. A higher level than normal suggests inflammation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 21 | 17
mg/L | 3.29 (6.85) | 1.4 (2.22)

7. Other Pre Specified Outcome: Characterization of the Immune System and Inflammation - WBC in CFS
Description: Blood and CSF were collected from healthy and ME/CFS participants at baseline. A comparison of the White Blood cell Count in Cerebrospinal Fluid (WBC in CFS), i.e., a measurement of the number of white blood cells in the cerebrospinal fluid, in the two populations is reported. Higher levels than normal suggest inflammation or infection in the central nervous system.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: number WBCs/uL
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 21 | 17
number WBCs/uL | 1.0 (1.124) | 1.313 (1.662)

8. Other Pre Specified Outcome: Mitochondrial Extracellular Flux Assay
Description: The oxygen consumption rate of peripheral blood mononuclear cells per unit of time when the cells are in their normal, unprovoked state of function measured in Basal (units) was measured in Healthy and ME/CFS participants at baseline. This is a standard measure of mitochondrial respiration that is responsible for providing energy to cells.
Time Frame: Baseline
Population: Technical issues with assay prevented complete dataset.
Measure: Median (Inter-Quartile Range); unit: Pmol/min
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 13 | 14
Pmol/min | 46.7 [26.2 to 58.0] | 52.1 [41.0 to 84.9]

9. Other Pre Specified Outcome: Effect of Maximal Exertion on Autonomic Function as Measured by SDNNi in Healthy and ME/CFS Participants.
Description: Variability of the time between heartbeats can be used to measure alterations in autonomic function. The Standard Deviation of the Normal-to-Normal Intervals (SDNNi) is a measure of the amount of beat to beat variability between each normal heartbeat collected over a 24 hour period. These results compare the SDNNi in healthy and ME/CFS participants at baseline.
Time Frame: Baseline
Population: Data from participants on cardiac medications were excluded.
Measure: Mean (Inter-Quartile Range); unit: ms
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 19 | 13
ms | 67.8 [58.9 to 77.1] | 56.3 [46.1 to 64.4]

10. Other Pre Specified Outcome: Clinical Response Effect of Tilt Table Testing
Description: Persons with autonomic dysfunction will often have symptoms provoked by having an up-to-40 minutes long tilt table test. The percentage of participants in each group having severe enough symptoms which required the test to be stopped in Healthy and ME/CFS participants at baseline.
Time Frame: Baseline
Population: Two participants were unable to complete due to technical difficulties with procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 19 | 17
percentage of participants | 36.8 | 58.8

11. Other Pre Specified Outcome: Characterization of the Pattern of Microbiome in Stool
Description: Stool samples were taken from Healthy and ME/CFS participants at baseline. The number of specific types of bacteria, using the Least Known Taxon (LTK) units, were measured with the Shotgun Metagenomic method.
Time Frame: Baseline
Population: Single batch analyzed on subset of participants
Measure: Mean (Standard Deviation); unit: LTK
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 17 | 15
LTK | 477 (32.9) | 427 (44.1)

12. Other Pre Specified Outcome: Test of Variables of Attention (TOVA)
Description: The TOVA is a measure of cognitive function that assesses attention and inhibitory control. The test is used to measure a number of variables involving the test taker's response to either a visual or auditory stimulus measured during a "simple, yet boring, computer game". These measurements are then compared to the measurements of a group of people without attention disorders who took the T.O.V.A. The range of values for the score, after normalization to the population, is -10 to +10, with a lower score representing a worse attention score. The test was administered to Healthy and ME/CFS participants at baseline.
Time Frame: Baseline
Population: Not all participants were able to complete test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 18 | 15
score on a scale | 1.1 (3.6) | 0.9 (4.7)

13. Other Pre Specified Outcome: Paced Auditory Serial Addition Test (PASAT)
Description: The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. Single digits are presented every 3 seconds and the patient must add each new digit to the one immediately prior to it. The test score is the total number of correct trials out of a possible 60. The test was administered to Healthy and ME/CFS participants at baseline.
Time Frame: Baseline
Population: Not all participants were able to complete test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
Number analyzed (Participants) | 17 | 15
score on a scale | 52.4 (12.1) | 52 (11)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Arm/Group | Healthy Volunteer Participants | ME/CFS Participants
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 14/25 | 23/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteer Participants (N=25) | ME/CFS Participants (N=27)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 12 (13)
Cerebrospinal fluid leakage (Nervous system disorders) | 6 (6) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 6 (12)
Headache (Nervous system disorders) | 3 (3) | 11 (15)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Movements Involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extremity pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Paresthesia (Nervous system disorders) | 2 (3) | 4 (4)
Pre-syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myaligia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02669212/Prot_SAP_000.pdf